CLINICAL TRIAL: NCT05872529
Title: Turkish Precision Anaesthesia Study Project
Acronym: TuPASProject
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University (Other)
Collaborators: Ankara University (Other); Marmara University (Other); Istanbul University - Cerrahpasa (Other); Acibadem University (Other); Cukurova University (Other); Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Özlem Korkmaz Dilmen, Prof MD, Istanbul University - Cerrahpasa
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Screening
Other Study IDs: IREANET001
Record Dates: First submitted 2023-05-03; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Delirium; Neurocognitive Disorders
Keywords: Delirium; Neurocognitive Disorders; electroencephalography; Postoperative
MeSH Terms: conditions — Delirium; Neurocognitive Disorders | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Before and After model
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BEFORE (No Intervention): The incidence of the POD and PND will determine before the education which consists processed EEG monitoring and SBI approach
- AFTER (Active Comparator): The incidence of the POD and PND will determine after the education which consists processed EEG monitoring and SBI approach
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — The education which consists processed EEG monitoring and SBI approach
  Arms: AFTER

SUMMARY:
Postoperative delirium (POD) and postoperative neurocognitive disorder (PND) increase the length of hospital stay, morbidity and mortality, especially in elderly patients. Although several risk factors were determined and incidence trials were performed on the development of POD and PND, there has not yet been a multicentre, large-participant study in Turkish population. The SBI approach monitor, detect and help physicians and all perioperative team members to decrease and avoid the adverse side effects of surgery and anaesthesia. In this "before and after" design trial the incidence of POD and PND will be compared before and after education which consists processed EEG and SBI approach.

The primary aim of the study is to determine the effect of education which consists processed EEG monitoring and regularly assessment of patient's stress, anxiety, pain, nausea, vomiting, thirst, hunger and better communication at the pre- and postoperative period on the incidence of POD. The secondary aim of the study is to assess the effect of the Safe Brain Initiative approach on patients' thirst feeling, stress-anxiety levels, postoperative pain, postoperative nausea and vomiting, well-being, satisfaction, length of PACU or recovery room stay, length of hospital stay, incidence of PND and in hospital and 3-month mortality. Also, the physicians', nurses' and patients satisfaction will be assessed.

DETAILED DESCRIPTION:
Postoperative delirium (POD) and postoperative neurocognitive disorder (PND) increase the length of hospital stay, morbidity and mortality, especially in elderly patients. Although several risk factors were determined and incidence trials were performed on the development of POD and PND, there has not yet been a multicentre, large-participant study in Turkish population. The EJA guideline recommends depth of anaesthesia monitoring, especially in frail patients since intraoperative burst suppression increases the risk of PND. American guideline emphasizes that the effect of processed EEG monitoring on POD cannot be fully demonstrated, but it may reduce PND. Yet, processed EEG monitors, when simplified to an index number, may not accurately reflect the depth of anaesthesia. To detect vulnerable patients, EEG training can be easily implemented. Thus, the incidence of POD and PND may decrease.

Additionally, not just EEG monitoring but also regular assessment of patients' stress, anxiety, pain, nausea, vomiting, thirst, and hunger during the pre-and postoperative period and better communication with the patients would reduce the risk of POD. That's why we will use the Safe Brain Initiative (SBI) approach. The SBI approach monitor, detect and help physicians and all perioperative team members to decrease and avoid the adverse side effects of surgery and anaesthesia. In this "before and after" design trial the incidence of POD and PND will be compared before and after education which consists processed EEG and SBI approach.

The primary aim of the study is to determine the effect of education which consists processed EEG monitoring and regularly assessment of patient's stress, anxiety, pain, nausea, vomiting, thirst, hunger and better communication at the pre- and postoperative period on the incidence of POD. The secondary aim of the study is to assess the effect of the Safe Brain Initiative approach on patients' thirst feeling, stress-anxiety levels, postoperative pain, postoperative nausea and vomiting, well-being, satisfaction, length of PACU or recovery room stay, length of hospital stay, incidence of PND and in hospital and 3-month mortality. Also, the physicians', nurses' and patients satisfaction will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients who will scheduled for non-cardiac, non-cranial surgery under general anaesthesia
* Patients who will undergo intraoperative processed EEG monitoring

Exclusion Criteria:

* Patients who will undergo outpatient, cardiac or intracranial surgery
* Patients undergoing surgery with regional anesthesia
* Alzheimer disease
* Psychiatric disorder
* Using antipsychotic drug
* Who will refuse to participate in study w
* Who scheduled for a second surgery within 3 months
* Who admitted to the ICU postoperatively with intubated and sedated

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2200 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative delirium | Up to postoperative 3 days
  POD will be assessed by Nu-DESC

SECONDARY OUTCOMES:
The incidence of postoperative neurocognitive disorder | Postoperative Month 3
  PND will be assessed by WHODAS2

OTHER OUTCOMES:
Duration of recovery room stay | 24 hours
  Duration of recovery room stay will be recorded
Duration of hospital stay | 2 weeks
  Duration of hospital stay will be recorded
Mortality | Postoperative Month 3
  Mortality will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Korkmaz Dilmen, Prof, Principal Investigator — Istanbul University- Cerrahpasa, Cerrahpasa Medical Faculty; Basak Ceyda Meco, Prof, Principal Investigator — Ankara University, Department of Anesthesiology and Intensive Care
Locations (1):
- Istanbul University - Cerrahpasa, Department of Neurosurgery, Neurosurgical Theaters, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sumner M, Deng C, Evered L, Frampton C, Leslie K, Short T, Campbell D. Processed electroencephalography-guided general anaesthesia to reduce postoperative delirium: a systematic review and meta-analysis. Br J Anaesth. 2023 Feb;130(2):e243-e253. doi: 10.1016/j.bja.2022.01.006. Epub 2022 Feb 17. PMID 35183345
- [Result] Evered L, Silbert B, Knopman DS, Scott DA, DeKosky ST, Rasmussen LS, Oh ES, Crosby G, Berger M, Eckenhoff RG; Nomenclature Consensus Working Group. Recommendations for the nomenclature of cognitive change associated with anaesthesia and surgery-2018. Br J Anaesth. 2018 Nov;121(5):1005-1012. doi: 10.1016/j.bja.2017.11.087. Epub 2018 Jun 15. PMID 30336844
- [Result] Kong H, Xu LM, Wang DX. Perioperative neurocognitive disorders: A narrative review focusing on diagnosis, prevention, and treatment. CNS Neurosci Ther. 2022 Aug;28(8):1147-1167. doi: 10.1111/cns.13873. Epub 2022 Jun 1. PMID 35652170
- [Result] Radtke FM, Franck M, Lendner J, Kruger S, Wernecke KD, Spies CD. Monitoring depth of anaesthesia in a randomized trial decreases the rate of postoperative delirium but not postoperative cognitive dysfunction. Br J Anaesth. 2013 Jun;110 Suppl 1:i98-105. doi: 10.1093/bja/aet055. Epub 2013 Mar 28. PMID 23539235